CLINICAL TRIAL: NCT04967274
Title: Contributions of the Reticulospinal System to Movement Control and Functional Recovery in Patients With Spinal Cord Injury
Brief Title: Reticulospinal Control of Movements
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2021-00973
Record Dates: First submitted 2021-05-26; First posted 2021-07-19 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Spinal Cord Injuries; Healthy
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: Each participants receives real and control interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Spinal cord injured subjects (Experimental)
  Interventions: Procedure: Startling acoustic stimulus

INTERVENTIONS:
Procedure: Startling acoustic stimulus — StartReact: involuntary triggering of a planed movement by a loud acoustic stimulus (Transcranial magnetic stimulation).

SUMMARY:
Accurate movement execution is a result of a complex interplay between various muscle groups whose activity is controlled by different areas of the central nervous system. Besides the corticospinal system, the phylogenetically old reticulospinal system is a key motor system controlling different elementary movements including posture, locomotion and reaching across all mammals. In contrast to the extensively investigated corticospinal system, there is only sparse knowledge on the motor physiology of the functionally important reticulospinal system in humans. Reticulospinal motor control can be assessed with the StartReact paradigm which is based on the activation of reticulospinal motor circuitries by startling acoustic stimuli. The StartReact phenomenon is characterized by a shortening in movement reaction time which is mediated by a startle-triggered, early release of a planned motor program by the reticulospinal system. Thus, StartReact is a unique tool to examine reticulospinal involvement on human motor control under physiological and pathological conditions. StartReact assessments will be supplemented by comprehensive 3-D kinematic analysis and muscle activity recordings (i.e. electromyography) to gain quantitative insights into reticulospinal movement control.

The first objective of this clinical study is to gain more insights into the mechanisms underlying StartReact and to advance the knowledge on reticulo-spinal motor physiology regarding different movement tasks (i.e. simple single-joint movements, complex multi-joint movements and bilateral hand movements) in healthy subjects. The findings of these experiments will provide new insights into proximal-distal, flexor-extensor and upper-lower extremity gradients in reticulospinal motor control of healthy subjects. Moreover, the results will expand the StartReact paradigm to complex, functionally more relevant movements (i.e. reaching and stepping tasks requiring endpoint accuracy; co-operative, bilateral hand movements) for which the involvement of the reticulo-spinal system is not yet understood.

The second goal of this project is to use the StartReact paradigm to shed more light onto the role of reticulospinal plasticity in functional recovery of patients with spinal cord injury (SCI). Whereas preclinical findings emphasize a remarkable potential of the reticulospinal system for neuroplastic adaptations underlying functional recovery, there is only little evidence from clinical trials in the field of SCI. First, the study aims at monitoring StartReact effects in hand and leg muscles of patients with acute SCI over a period of 6 months. Simultaneous tracking of StartReact effects and motor recovery will allow to closely relate processes of reticulospinal plasticity to functional recovery in patients with acute SCI. Second, the focus will be on the re-weighting of descending motor control (i.e. cortico- vs. reticulospinal system) in response to SCI and investigate the distinct contributions of the cortico- and reticulospinal system to motor recovery in patients with chronic SCI.

The findings of this project will advance the mechanistic understanding on the motor physiology and neurorestorative capacity of the reticulospinal system in humans. New insights from these projects will hopefully translate into a better exploitation of this important motor system in clinical trials that aim to improve motor recovery in patients with SCI.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent as documented by signature

For SCI patients:

* ASIA Impairment scale (AIS) A-D
* Focal damage at cervical (C4-C7; i.e. damage rostral of the spi-nal segments innervating the examined hand and leg muscles) or thoracic (T4-T12; i.e. damage caudal of the spinal segments innervating the m. abductor digiti minimi, but rostral of the spi-nal segments innervating the m. tibialis anterior)
* Patients with cervical SCI must reveal bilaterally intact ulnar nerves as demonstrated by normal compound motor action potential (cMAP), nerve conduction velocity (NCV) and F-wave latencies in clinical neurography.
* Patients with thoracic SCI must reveal bilaterally intact tibial and peroneal nerves as demonstrated by normal cMAP, NCV and F-wave latencies

Exclusion Criteria:

* Women who are pregnant or breast feeding
* Current neurological problems other than SCI and related impairments
* Current orthopaedic problems affecting upper and lower extremity movements
* History of alcohol abuse or the intake of psychotropic drugs
* History of major cardiac condition (e.g., infarction, insufficiency (NYHA II-IV))
* History of major pulmonary condition (e.g., chronic obstructive pulmonary disease (GOLD II-IV))
* Current major depression or psychosis
* Fever of unknown origin

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2022-01-15 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
EMG analysis (i.e. shortening of movement reaction time of target muscle(s)) during Loud vs. Moderate Acoustic Stimuli (LAS vs. MAS) | Baseline
Change in EMG analysis (i.e. shortening of movement reaction time of target muscle(s)) | Change in shortening of movement reaction time between baseline and visit 1 (7-14 days).
Change in EMG analysis (i.e. shortening of movement reaction time of target muscle(s)) | Change in shortening of movement reaction time at 3 and 6 months relative to baseline.
Intramuscular coherence of paired EMG signals of the tibialis anterior muscle to assess corticospinal drive in the StartReact paradigm. | Baseline
Modulation of EMG reflex responses (as induced by electrical ulnar nerve stimulation) by simultaneous acoustic stimulation with LAS | Baseline
Transcranial magnetic stimulation (TMS) to investigate corticospinal physiology/ integrity. | Baseline

SECONDARY OUTCOMES:
Analysis of movement patterns of fast vs. slow movements based on 3D kinematics. | Baseline
Endpoint accuracy of fast vs. slow reaching and stepping movements based on a combined Virtual Reality (VR)/ kinematic system. | Baseline
Graded Redefined Assessment of Strength, Sensibility, and Prehension (GRASSP) to measure upper extremity function (only for SCI) | The outcome is used for 2 sub-projects of this study: one sub-project conducts GRASSP at > 12 months after spinal cord injury, whereas the other sub-project conducts GRASSP at 3 visits (at < 1, 3 and 6 months after spinal cord injury).
International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) (only for SCI) | The outcome is used for 2 sub-projects of this study: one sub-project conducts ISNCSCI at > 12 months after spinal cord injury, whereas the other sub-project conducts ISNCSCI at 3 visits (at < 1, 3 and 6 months after spinal cord injury).
10-meter walk test (only for SCI) | Baseline
6-minute walk test (only for SCI) | Baseline
Modified Ashworth Scale (MAS) (only for SCI) | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Freund, Prof. Dr., Principal Investigator — University of Zurich
Locations (1):
- Balgrist University Hospital, Zurich, Switzerland